CLINICAL TRIAL: NCT06071910
Title: Emergency Resuscitative Endovascular Balloon Occlusion of the Aorta in Out of Hospital Cardiac Arrest
Acronym: ERICA-ARREST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: East Anglian Air Ambulance (Unknown); Rosetrees Trust (Other); The Dowager Countess Eleanor Peel Trust (Unknown); The Drummond Foundation (Unknown)
Responsible Party: Principal Investigator, Paul Rees, Principal Investigator, Queen Mary University of London
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 296654
Record Dates: First submitted 2023-07-14; First posted 2023-10-10 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Cardiac Arrest; Cardiac Arrhythmia; Ventricular Fibrillation; Ventricular Arrythmia; Pulseless Electrical Activity
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest; Arrhythmias, Cardiac; Ventricular Fibrillation

STUDY DESIGN:
Intervention Model Description: Sequential patients with OHCA in air ambulance operational area
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Aortic balloon occulsion (Other): Delivery of ER-REBOA catheter to achieve aortic occlusion during resuscitation for out of hospital cardiac arrest, refractory to conventional advanced life support
  Interventions: Device: ER-REBOA catheter

INTERVENTIONS:
Device: ER-REBOA catheter — To achieve rapid aortic occlusion
  Other Names: Aortic balloon occlusion; REBOA

SUMMARY:
This study will assess the feasibility of performing pre-hospital resuscitative endovascular balloon occlusion of the aorta (REBOA) as an adjunct to conventional Advanced Life Support (ALS) in patients suffering from non-traumatic out of hospital cardiac arrest (OHCA). As well as providing valuable insights into the technical feasibility of performing this procedure as part of a resuscitation attempt, the study will also document the beneficial physiological effects of REBOA in this group of patients.

DETAILED DESCRIPTION:
This study will assess the feasibility of performing pre-hospital resuscitative endovascular balloon occlusion of the aorta (REBOA) as an adjunct to conventional Advanced Life Support (ALS) in patients suffering from non-traumatic out of hospital cardiac arrest (OHCA). As well as providing valuable insights into the technical feasibility of performing this procedure as part of a resuscitation attempt, the study will also evaluate the physiological benefits of REBOA in this group of patients.Twenty patients will be enrolled in this study. The protocol is designed according to the IDEAL framework Stage 2a1 for evaluating surgical interventions, where a small prospective case series is used to test and stabilise the intervention. The study will help establish whether the technique is ready for evaluation in a prospective multi-centre randomised study.

Background

In England, the average overall survival to hospital discharge from Emergency Medical Service (EMS) treated OHCA is 8.6%. This is significantly lower than in other European, Scandinavian and North American settings, where survival rates range from 14-21%.

Improving survival rates from OHCA is a major priority for the Resuscitation Council (UK), the British Heart Foundation and National Health Service (NHS) England and was identified as a key area for improvement by the Department of Health. The most common cause of sudden OHCA is coronary artery disease.

The current goals for pre-hospital management of OHCA are to provide early effective CPR to provide brain and heart blood flow, early defibrillation to restart the heart, and to support the circulation with advanced life support once available. Minimising periods of "no-flow" or "low-flow" are key to setting the conditions for successful resuscitation, and avoiding irreversible damage to critical organs, in particular the brain.

Other adjuncts to Advanced Life Support

Other therapeutic modalities such as percutaneous coronary intervention (PCI) and thrombolysis are well-documented therapies included in current ALS guidelines, but these require the patient to have a stable return of spontaneous circulation, and they can only realistically be provided after the patient has been fully resuscitated and delivered to a hospital. Even where this is possible, when these treatments are provided during ongoing CPR they are usually futile. Extracorporeal membrane oxygenation (ECMO) CPR (ECPR - the provision of an emergency heart-lung bypass circuit) is a suggested intervention for patients in refractory cardiac arrest with encouraging data from some observational studies. However, ECPR is a complex intervention that requires considerable resources and training. It is not currently available in the majority of UK hospitals. No prehospital services can currently deliver ECPR, a situation which is likely to persist. A capability gap exists which this study aims to address.

Pre-Hospital REBOA: anticipated clinical benefits and challenges

REBOA is a technique used to provide temporary occlusion of the aorta by inflation of an intra-aortic balloon. REBOA has been used to manage haemorrhagic shock and traumatic cardiac arrest by controlling bleeding and allowing a patient's physiology to stabilize.

REBOA has been proposed as an adjunct treatment in managing non-traumatic cardiac arrest patients. Thoracic aortic occlusion with a balloon provides a redistribution of the cardiac output to organs proximal to the occlusion. The resultant effect increases the coronary perfusion pressure (CPP); the driving force of blood through the coronary arteries. CPP is calculated as the diastolic aortic pressure minus the right atrial pressure: higher aortic diastolic blood pressure results in higher coronary perfusion pressure. REBOA during resuscitation also increases blood flow to the carotid arteries, cerebral arteries and cerebral perfusion pressure. This improves blood flow to the brain, which may protect it from damage.

During cardiac arrest, brain tissue is especially susceptible to hypoxemia; improved peri-resuscitation blood pressure may improve brain perfusion. Cerebral oximetry, which measures regional cerebral oxygen saturation (rSO2) by near-infrared spectroscopy, has emerged as a potentially helpful marker of cerebral ischaemia during CPR. In preclinical and clinical studies, higher rSO2 values during CPR are associated with improved cardiac arrest survival and neurologic outcome. rSO2 could be used as a surrogate marker for cerebral perfusion.

It is anticipated that REBOA can improve the perfusion of the brain and heart during CPR. Moreover, improved aortic blood pressure will have the potential clinical benefit of improving rates of ROSC. REBOA could also provide bridging therapy for patients who are refractory to conventional CPR until the patient is transferred to a unit capable of providing ECPR. Thus, REBOA could equally offer a "bridge to ROSC" or a "bridge to ECPR" in suitable patients.

Preclinical data

Animal data confirm multiple haemodynamic and electrophysiological benefits to aortic balloon occlusion during cardiopulmonary resuscitation. In 1993, Tang et al used a porcine model of cardiac arrest to investigate the effects of aortic balloon occlusion during resuscitation of twenty anaesthetised, ventilated pigs. After inducing ventricular fibrillation, chest compressions were commenced, and the animals randomised to various intervention arms, including aortic balloon occlusion by means of a 10 French (F) device inserted via the left femoral artery. This study demonstrated that the efficacy of CPR was augmented by balloon occlusion, resulting in better coronary perfusion pressure, and strikingly improved both the likelihood of successful resuscitation and 48 hour survival compared with control groups.

Building on their previous animal studies showing improvements in coronary perfusion pressure associated with an endovascular resuscitation technique, in 1996 a US group led by Manning combined aortic balloon occlusion with retrograde aortic perfusion in a canine model of cardiac arrest. Eight dogs (including 4 control animals) were sedated, intubated, catheterized, and instrumented to record ECG, right atrial pressure, and aortic pressure during resuscitation after ventricular fibrillation (VF) induced cardiac arrest. After 10 minutes of VF-induced arrest, mechanical CPR was initiated. 2 minutes later, the 4 study animals received selective aortic arch perfusion (SAAP - a combination of aortic occlusion and retrograde aortic perfusion). Defibrillation was attempted after 3 minutes of CPR and every minute thereafter. Animals received standard-dose epinephrine every 3 minutes by means of an intra-aortic catheter. SAAP infusion resulted in significant increases in median frequency and peak amplitude of VF in the SAAP group compared with the control group, coupled with an improvement in coronary perfusion pressure. This method of resuscitation was reliable in allowing restoration of a stable perfusing rhythm after defibrillation. The authors comment that the changes in peak amplitude and median frequency of the underlying cardiac rhythm, induced by improved coronary perfusion during resuscitation were likely responsible for the increased likelihood of successful defibrillation.

Gedeborg and colleagues further investigated the role of aortic balloon occlusion in order to evaluate the effects of this intervention on haemodynamics and the frequency of restoration of spontaneous circulation. Ventricular fibrillation was induced in 39 anaesthetised piglets, followed by an 8-min non-intervention interval. In a haemodynamic study (n = 10), closed chest CPR was performed for 7 min before an intra-aortic balloon was inflated. This intervention increased mean arterial blood pressure by 20% and increased coronary artery blood flow by 86%. Common carotid artery blood flow also increased by 62%. All these changes were statistically significant. Interestingly, although administration of epinephrine further increased mean arterial blood pressure and coronary artery blood flow, a paradoxical decrease was seen in common carotid artery blood. In a study of short-term survival, nine out of 13 animals (69%) in the balloon group and in three out of 13 animals (23%) in the control group had spontaneous circulation restored.

In 2002, Sesma et al compared the effectiveness of CPR with and without balloon aortic occlusion balloon, monitoring capnography, coronary and cerebral perfusion pressure (CePP) in normothermic induced VF arrest in a crossover study of 14 pigs. Aortic balloon deployment resulted in significant circulatory improvements: End-tidal carbon dioxide (ETCO2) rose by 38%, and coronary perfusion pressure rose initially from 10 to 29 mm Hg - an increase of 150%. The CePP improved from 12 to 39 mm Hg after the balloon was inflated, representing an increase of 200%. In all cases, the differences were statistically significant (P < .0001), although they diminished as the resuscitation progressed in time.

Most recently, Hutin's resuscitation research group in Paris reported on the use of REBOA as a potential alternative to epinephrine in the management of non-traumatic cardiac arrest, assessing the comparative effects of epinephrine vs. REBOA on ROSC, haemodynamics and cerebral circulation in a porcine model of cardiac arrest. After 4 min of cardiac arrest and 18 min of basic life support (BLS) using a mechanical CPR device, animals were randomised to receive either REBOA or epinephrine administration before defibrillation attempts. Six animals were included in each experimental arm. Haemodynamic parameters were similar in both groups during BLS. After epinephrine administration or REBOA, mean arterial pressure, coronary and cerebral perfusion pressures similarly increased in both groups. However, carotid blood flow (CBF) and cerebral regional oxygenation saturation were significantly higher with REBOA as compared to epinephrine administration (+ 125% and + 40%, respectively). ROSC was obtained in 5 animals in both groups. After resuscitation, CBF remained lower in the epinephrine group as compared to REBOA. This study confirms the beneficial haemodynamic effects of aortic balloon occlusion during cardiac arrest, and hints at a potential role in reducing the deleterious effects of bolus epinephrine on the cerebral circulation. This is in accordance with Gedeborg's findings with respect to post-epinephrine carotid flow.

Clinical data

Human data concerning the potential role of aortic balloon occlusion include a number of case reports of the use of transient aortic occlusion during refractory cardiac arrest in the setting of the cardiac catheter lab or cardiac operating theatre. Deakin and Barron describe two cases of severe haemodynamic instability and intermittent cardiac arrest where aortic balloon occlusion was used: In the first case, mean radial artery pressure rose from 71/14 mmHg (mean=33 mmHg) to 92/24 mmHg (mean=47 mmHg). In the second case, mean radial artery pressure rose from 48/21 mmHg (mean=25 mmHg) to 62/26 mmHg (mean=36 mmHg). Calculated coronary artery perfusion pressure in case 1 increased from -2 to 8 mmHg, and in case 2 increased from 15 to 18 mmHg, suggesting that occlusion of the descending aorta during cardiac massage may improve coronary and cerebral perfusion pressures.

Aslanger et al report on a patient with myocardial infarction and severe multivessel coronary artery disease undergoing coronary angiography who suffered severe hypotension during the procedure. Despite inotropic support, cardiac arrest ensued. CPR was initiated and advanced life support (ALS) was performed according to guidelines. A peak blood pressure of approximately 100 mmHg was observed during chest compressions. There were no arterial waveforms on the monitor between chest compressions throughout this period, and asystole developed. During ongoing CPR, the 7F femoral access sheath was exchanged for an 8F femoral intraaortic catheter sheath. A 40-ml intraaortic balloon catheter was delivered and inflated. Complete occlusion of the descending aorta was confirmed by loss of the arterial waveform from the femoral sheath side-port during chest compressions. Thirty seconds after balloon occlusion, spontaneous gasping appeared. Forty-five seconds after balloon occlusion, a heartbeat of 35 bpm was observed. This rhythm accelerated progressively, and sinus rhythm was restored after a minute. A pulse check confirmed a strong carotid pulse. At this point, the balloon was deflated to terminate aortic occlusion and the blood pressure monitored from the femoral sheath increased to 80/50 mmHg. An intraaortic balloon catheter was attached to an intraaortic pump console and standard counterpulsation was started along with a dopamine infusion. During 12 h of follow up, the systolic arterial blood pressure was about 110 mmHg and the dopamine dose was weaned down. After the patient had regained consciousness, she was extubated and all mechanical and inotropic support was stopped. The following day, the patient's clinical status was excellent and the overall performance category (OPC) and cerebral performance category (CPC) scores were both one. The authors comment that their inability to document coronary perfusion pressure is a limitation of this case report. The suggest, however, that resumption of breathing and ROSC were valid surrogates for improved cerebral and coronary perfusion respectively, and it seems likely that this improvement was solely due to timely aortic balloon deployment in the context of refractory cardiac arrest despite guideline-directed resuscitation.

A similar case is reported by a group at Barts Heart Centre (Kalogeropoulos et al); mechanical CPR was combined with intermittent aortic balloon counterpulsation (IABP) in a 49 year old male who suffered on-table cardiac arrest during emergency percutaneous coronary intervention for acute myocardial infarction. Although this case differs as the intraaortic balloon device allowed rapid, synchronised inflation and deflation of the aortic balloon (this preventing downstream organ ischaemia and offering additional left ventricular unloading), the authors suggest IABP could be considered as an adjunctive intervention to mechanical CPR (mCPR) to enhance myocardial perfusion and expedite and facilitate ROSC. Furthermore, in centres without availability of more advanced mechanical support (such as Impella or ECMO devices), IABP as a bailout adjunctive therapy to mCPR might contribute to improvement of myocardial perfusion and central hemodynamic parameters and shorten the time to ROSC, allowing successful bridging to more advanced mechanical circulatory support (MCS) modalities, transfer to a PCI-capable center, and successful revascularization. In this case, ROSC was achieved and, after a prolonged hospital stay, the patient made a full recovery and was neurologically intact.

The use of a REBOA device as an adjunct to resuscitation of patients has been described in Italy by Gamberini and colleagues, in a mixed cohort of traumatic and non-traumatic cardiac arrests. The procedure was performed using one of two different aortic balloon systems by critical care physicians operating within hospital or alongside emergency medical service teams at the scene. Of the 18 successful reported REBOA procedures, 11 were performed in non-traumatic OHCA patients (7 in-hospital and 4 prehospital) with a median age of 52 years; the most common suspected aetiology was cardiac disease (5/11), while other causes were: massive pulmonary embolism, hyperkalaemia, a neurological syndrome and cardiac tamponade. In 8/11 cases, balloon inflation caused led to a measurable increase in ETCO2 equal or higher than 10 mmHg at one minute after occlusion and median etCO2 increased from 15 to 24 mmHg (p = 0.016). The majority of patients experiencing an increase in etCO2 equal or higher than 10 mmHg at one minute after occlusion also got transient ROSC. However, a sustained ROSC (lasting over 20 min) was achieved by only 4 out of the 11 patients. In the absence of measured haemodynamic variables, an increased in ETCO2 possibly represents a surrogate for enhanced circulation during ongoing CPR compared with baseline.

The most comprehensive feasibility study of REBOA in nontraumatic cardiac arrest was performed by Norwegian helicopter emergency medical services (HEMS) and reported in 2019 by Brede et al. A safety monitoring programme ran alongside this prospective observational feasibility study to ensure that the interventional procedure itself did not adversely affect the quality of advanced cardiac life support. 10 patients received REBOA, delivered at-scene by the HEMS physician, in a cohort of patients with a mean age of 63 years (range 50-74 years). REBOA procedure was successful in all cases, with 80% success rate on first attempt. This is likely to be due to the design of an effective and intensive team-based training programme. Mean procedural time was 11.7 minutes (SD 3.2, range 8-16). Mean end-tidal CO2 increased by 1.75 kiloPascals (kPa) after 60 seconds compared with baseline (P<0.001). Six patients achieved return of spontaneous circulation (60%), 3 patients survived to reach hospital admission, and 1 patient survived past 30 days. The safety-monitoring program identified no negative influence on the advanced cardiac life support quality. The significant increase in end-tidal CO2 after occlusion suggests improved organ circulation during cardiopulmonary resuscitation. Of note, this patient cohort were quite advanced in terms of the delay of the HEMS team in reaching the incident location, probably reflecting long travel times due to geographical distance. Despite short procedural times (mean time from arrival at scene to REBOA deployment was 11.7±3.2 mins, emergency call to scene times were 45.6±6.3 minutes. This means that REBOA was applied 75.3 minutes after the onset of cardiac arrest. It is certainly possible that the positive response to REBOA might be more pronounced (and thus more likely to lead to ROSC) where it is applied earlier during the cardiac arrest; perhaps after the 20 minute point, which is suggested as the point of inflexion at which conventional ALS should be deprioritised in favour of novel therapies such as ECMO-CPR, where they are available.

Rationale

Use of REBOA as an adjunct treatment to ALS in non-traumatic cardiac arrest is a novel treatment which has potential to improve outcomes in a patient group who currently experience dismal rates of death and neurological disability. This study will test the feasibility of deploying REBOA in a UK prehospital critical care team. It is not a trial to test a medical device or to compare outcomes between different treatments.

No UK prehospital care services are currently able to deploy REBOA in the setting of OHCA. However, as outlined in the previous sections, there is good physiological data to support its potential use as a bridge to ROSC. In this setting, REBOA could be expected to raise aortic diastolic blood pressure, increase coronary perfusion, and enhance cerebral perfusion. Potentially, these physiological improvements could enhance the chance of achieving ROSC, and preserve blood flow to the brain, improving the chances of surviving with preserved brain function.

Whilst a previous single-centre observational study has demonstrated the feasibility of REBOA in non-traumatic OHCA in Norway, this will be the first study of HEMS-team delivered REBOA for OHCA in the UK. Additionally, this study will document the physiological response to REBOA in the setting of ongoing resuscitation, which might underpin its future utility. This study will also aim to provide the intervention in a more rapid timescale. In the published datasets, due primarily to geographical constraints, there was a delay of 45 to 50 minutes from the time of emergency call to initiating establishing REBOA. It is likely to be a time-critical intervention, and the compressed geographical catchment area of the study population, alongside a well-established and clinically-governed pre-existing arterial access program, should facilitate more rapid delivery.

Feedback from the EAAA patient group showed strong support for the study, with the group supportive of an innovation with potential to improve survival after cardiac arrest and acknowledging that EAAA are in an excellent position to carry out the study.

The study will follow the IDEAL framework for evaluation of a surgical intervention, using the Stage 2a prospective series of a novel technique to assess the feasibility of the technique in the setting.This will help inform potential development of a multi-centre randomised controlled trial.

Risk/ benefits

This is an invasive and demanding intervention in a population who are critically ill as they are in cardiac arrest and have not responded to standard ALS. Risks and mitigation plans are detailed further in section 10 and include:

* Interruption to ALS
* Inadvertent misplacement of REBOA catheter
* Access site complications such as puncture site bleeding, bruising and minor arterial dissection
* Lower limb and organ ischemia
* Occlusion of carotid artery
* Increased bleeding
* Risk of infection
* Risk to study personnel

The following steps will control or mitigate these risks:

* The procedure will be carried out by a small number of experienced physicians at EAAA who are already expert at ultrasound-guided femoral access during ongoing resuscitation (over 100 cases already successfully and safely achieved).
* All participating personnel will take part in a structured training program and be certified before they can perform the procedure.
* The equipment is well known and already used in a range of indications and patients
* The equipment is small gauge, which limits the risk of local complications.
* Following each procedure, the performing physician will be interviewed to discuss any safety concerns.

The study is justified based on the anticipated clinical benefits outlined above and with robust procedures in place to minimise risk.

ELIGIBILITY:
Inclusion criteria

* Non-Traumatic OHCA in patients within the East of England area AND with a East Anglian Air Ambulance (EAAA) REBOA team in attendance
* Patients below or equal to 80yrs of age and above or equal to 18yrs of age, according to available information/estimate at scene
* No flow <10 mins from data available (i.e. total period in OHCA with no CPR)
* In cardiac arrest (with no sustained ROSC) on arrival of the EAAA REBOA team

Exclusion criteria

* Patients aged less than 18 or above 80 years
* Known terminal illness
* Multiple severe co-morbidities
* Traumatic Cardiac Arrest (TCA)
* Inability to deploy mechanical CPR (e.g. LUCAS Device)
* Pregnancy, obvious or suspected

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Device delivery | Within 1 hour of initiation
  The proportion of patients where Pre-Hospital Zone 1 REBOA for OHCA is achieved, with balloon inserted to 35 - 55 cm, proximal arterial blood pressure transduced and evidence of loss of distal invasive blood pressure trace during CPR confirming aortic occlusion.
Procedural timings | Within 1 hour of initiation
  Time taken to achieve REBOA for OHCA in mins
  * Time taken from start of the procedure (arterial catheterization) to balloon inflation in mins
  * Total duration of REBOA (inflation to final deflation) in mins
  * Time from arrival at scene to REBOA (balloon inflation) in mins
  * Time from 999 call to REBOA (balloon inflation) in mins

SECONDARY OUTCOMES:
Haemodynamic and oxygenation responses | Within 1 hour of initiation
  Change in aortic diastolic pressure in mmHg
  * Change in central venous pressure in mmHg
  * Change in calculated coronary perfusion pressure (where cannulated) (CPP) mmHg
  These hemodynamic end-points will be presented as a consecutive case series (continuous data plots per patient) and a descriptive summary for the whole cohort of absolute values and change in values between key time intervals: Pre-occlusion, During Occlusion, Post- Occlusion.
Near Infra-Red Spectrometry | Within 1 hour of initiation
  Change in brain regional oxygen saturation (rSO2) in %
  These cerebral oxygenation end-points will be presented as a consecutive case series (continuous data plots per patient) and a descriptive summary for the whole cohort of absolute values and change in values between key time intervals: Pre-occlusion, During Occlusion, Post- Occlusion.
End Tidal CO2 | Within 1 hour of initiation
  Change in ETCO2 in KPa
  These circulatory-surrogate end-points will be presented as a consecutive case series (continuous data plots per patient) and a descriptive summary for the whole cohort of absolute values and change in values between key time intervals: Pre-occlusion, During Occlusion, Post- Occlusion.

CONTACTS AND LOCATIONS:
Locations (1):
- East Anglian Air Ambulance, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moriwaki Y, Tahara Y, Kosuge T, Suzuki N. Etiology of out-of-hospital cardiac arrest diagnosed via detailed examinations including perimortem computed tomography. J Emerg Trauma Shock. 2013 Apr;6(2):87-94. doi: 10.4103/0974-2700.110752. PMID 23723616
- [Background] Yannopoulos D, Bartos J, Raveendran G, Walser E, Connett J, Murray TA, Collins G, Zhang L, Kalra R, Kosmopoulos M, John R, Shaffer A, Frascone RJ, Wesley K, Conterato M, Biros M, Tolar J, Aufderheide TP. Advanced reperfusion strategies for patients with out-of-hospital cardiac arrest and refractory ventricular fibrillation (ARREST): a phase 2, single centre, open-label, randomised controlled trial. Lancet. 2020 Dec 5;396(10265):1807-1816. doi: 10.1016/S0140-6736(20)32338-2. Epub 2020 Nov 13. PMID 33197396
- [Background] Osborn LA, Brenner ML, Prater SJ, Moore LJ. Resuscitative endovascular balloon occlusion of the aorta: current evidence. Open Access Emerg Med. 2019 Jan 14;11:29-38. doi: 10.2147/OAEM.S166087. eCollection 2019. PMID 30666171
- [Background] Lendrum R, Perkins Z, Chana M, Marsden M, Davenport R, Grier G, Sadek S, Davies G. Pre-hospital Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) for exsanguinating pelvic haemorrhage. Resuscitation. 2019 Feb;135:6-13. doi: 10.1016/j.resuscitation.2018.12.018. Epub 2018 Dec 27. PMID 30594600
- [Background] Levis A, Greif R, Hautz WE, Lehmann LE, Hunziker L, Fehr T, Haenggi M. Resuscitative endovascular balloon occlusion of the aorta (REBOA) during cardiopulmonary resuscitation: A pilot study. Resuscitation. 2020 Nov;156:27-34. doi: 10.1016/j.resuscitation.2020.08.118. Epub 2020 Aug 29. PMID 32866549
- [Background] Tang W, Weil MH, Noc M, Sun S, Gazmuri RJ, Bisera J. Augmented efficacy of external CPR by intermittent occlusion of the ascending aorta. Circulation. 1993 Oct;88(4 Pt 1):1916-21. doi: 10.1161/01.cir.88.4.1916. PMID 8403337
- [Background] Manning JE, Murphy CA Jr, Hertz CM, Perretta SG, Mueller RA, Norfleet EA. Selective aortic arch perfusion during cardiac arrest: a new resuscitation technique. Ann Emerg Med. 1992 Sep;21(9):1058-65. doi: 10.1016/s0196-0644(05)80645-6. PMID 1514716
- [Background] Gedeborg R, Rubertsson S, Wiklund L. Improved haemodynamics and restoration of spontaneous circulation with constant aortic occlusion during experimental cardiopulmonary resuscitation. Resuscitation. 1999 Apr-May;40(3):171-80. doi: 10.1016/s0300-9572(99)00021-0. PMID 10395400
- [Background] Sesma J, Labandeira J, Sara MJ, Espila JL, Arteche A, Saez MJ. Effect of intra-aortic occlusion balloon in external thoracic compressions during CPR in pigs. Am J Emerg Med. 2002 Sep;20(5):453-62. doi: 10.1053/ajem.2002.32627. PMID 12216044
- [Background] Hutin A, Levy Y, Lidouren F, Kohlhauer M, Carli P, Ghaleh B, Lamhaut L, Tissier R. Resuscitative endovascular balloon occlusion of the aorta vs epinephrine in the treatment of non-traumatic cardiac arrest in swine. Ann Intensive Care. 2021 May 17;11(1):81. doi: 10.1186/s13613-021-00871-z. PMID 34002305
- [Background] Deakin CD, Barron DJ. Haemodynamic effects of descending aortic occlusion during cardiopulmonary resuscitation. Resuscitation. 1996 Nov;33(1):49-52. doi: 10.1016/s0300-9572(96)00992-6. PMID 8959773
- [Background] Aslanger E, Golcuk E, Oflaz H, Yilmaz A, Mercanoglu F, Bugra Z, Umman B, Nisanci Y. Intraaortic balloon occlusion during refractory cardiac arrest. A case report. Resuscitation. 2009 Feb;80(2):281-3. doi: 10.1016/j.resuscitation.2008.10.017. Epub 2008 Dec 6. PMID 19058900
- [Background] Kalogeropoulos AS, Kennon S, Karamasis GV, Smith EJ, Rees P. Successful Primary Percutaneous Coronary Intervention for Acute Myocardial Infarction During Resuscitation From Cardiac Arrest by Combined Mechanical Chest Compressions and Intra-aortic Balloon Pump Counterpulsation: A Case Report. A A Pract. 2018 Jun 15;10(12):323-326. doi: 10.1213/XAA.0000000000000707. PMID 29634573
- [Background] Gamberini L, Coniglio C, Lupi C, Tartaglione M, Mazzoli CA, Baldazzi M, Cecchi A, Ferri E, Chiarini V, Semeraro F, Gordini G; collaborators. Resuscitative endovascular occlusion of the aorta (REBOA) for refractory out of hospital cardiac arrest. An Utstein-based case series. Resuscitation. 2021 Aug;165:161-169. doi: 10.1016/j.resuscitation.2021.05.019. Epub 2021 Jun 3. PMID 34089774
- [Background] Brede JR, Lafrenz T, Klepstad P, Skjaerseth EA, Nordseth T, Sovik E, Kruger AJ. Feasibility of Pre-Hospital Resuscitative Endovascular Balloon Occlusion of the Aorta in Non-Traumatic Out-of-Hospital Cardiac Arrest. J Am Heart Assoc. 2019 Nov 19;8(22):e014394. doi: 10.1161/JAHA.119.014394. Epub 2019 Nov 11. PMID 31707942
- [Derived] Aziz S, Barratt J, Wilson-Baig N, Lachowycz K, Major R, Barnard EBG, Rees P. A protocol for the ERICA-ARREST feasibility study of Emergency Resuscitative Endovascular Balloon occlusion of the Aorta in Out-of-Hospital Cardiac Arrest. Resusc Plus. 2024 Jun 13;19:100688. doi: 10.1016/j.resplu.2024.100688. eCollection 2024 Sep. PMID 38974930
- See also: Consensus Paper on Out-of-Hospital Cardiac Arrest in England — https://www.resus.org.uk/sites/default/files/2020-05/OHCA_consensus_paper.pdf
- See also: Department of Health Cardiovascular Disease Team. Cardiovascular Disease Outcomes Strategy- Improving outcomes for people with or at risk of cardiovascular disease — https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment_data/file/217118/9387-2900853-CVD-Outcomes_web1.pdf